CLINICAL TRIAL: NCT04079335
Title: A Prospective Longitudinal Study of Fecal Microbiome and Calprotectin to Predict Relapse in Patients With Inflammatory Bowel Disease
Brief Title: A Prospective Longitudinal Study of Fecal Microbiome and Calprotectin to Predict Relapse in Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Profressor, Chinese University of Hong Kong
Other Study IDs: IBD MiREL
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic idiopathic inflammatory condition of the intestine, which results in diarrhea, rectal bleeding, urgency, weight loss and abdominal pain. The natural course of IBD is characterized by activity outbreaks and periods of remission. In most cases, relapses in Crohn's disease (CD) and in ulcerative colitis (UC) are unpredictable and despite effective medical treatment, a degree of subclinical inflammation may persist in the bowel wall, contributing to a significant risk of relapse.

In IBD, altered fecal microbiota signatures have been consistently reported which included a reduction in biodiversity with lower proportions of Firmicutes and increases in Proteobacteria and Bacteroidetes phylum members.

It is however unclear whether changes in microbial profile including diversity and composition can predict disease relapse in IBD. We hypothesize that fecal microbial signatures in conjunction with fecal calprotectin may play a role in predicting relapse in IBD patients.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic idiopathic inflammatory condition of the intestine, which results in diarrhea, rectal bleeding, urgency, weight loss and abdominal pain. The natural course of IBD is characterized by activity outbreaks and periods of remission. In most cases, relapses in Crohn's disease (CD) and in ulcerative colitis (UC) are unpredictable and despite effective medical treatment, a degree of subclinical inflammation may persist in the bowel wall, contributing to a significant risk of relapse.

Endoscopy has been used to monitor a disease but it is time-consuming, costly, invasive, and associated with certain risks of morbidity. Many patients are reluctant to undergo repeated endoscopic examinations, particularly when their disease is quiescent. Acute phase reactants have been used but their sensitivity and specificity in correlating to intestinal inflammatory activity are very low, and their capacity to predict disease relapse is poor and controversial. A number of fecal biomarkers have been evaluated for their utility for monitoring and predicting relapse in IBD but some of these biomarkers are also not specific.

In IBD, altered fecal microbiota signatures have been consistently reported which included a reduction in biodiversity with lower proportions of Firmicutes and increases in Proteobacteria and Bacteroidetes phylum members. In addition, disease remission and relapse are associated with microbial changes in both mucosal and fecal samples. In particular, a loss of species richness in Crohn's disease has been widely observed. Recently microbial biomarkers may differentiate between CD and UC. Furthermore, different microbial groups are associated with smoking habit and localization of the disease in CD and UC. It is however unclear whether changes in microbial profile including diversity and composition can predict disease relapse in IBD. We hypothesize that fecal microbial signatures in conjunction with fecal calprotectin may play a role in predicting relapse in IBD patients.

ELIGIBILITY:
Inclusion Criteria:

Patient with Crohn's Disease

1. Aged ≥18 years old
2. Confirmed diagnosis of ileo-colonic Crohn's disease according to established clinical, endoscopic and histologic criteria
3. History of at least one flare with symptoms that required intervention within 24 months before screening
4. Stable doses of immunosuppressive agents for at least 3 months if these agents are required
5. In clinical remission for at least 3 months, defined as Harvey Bradshaw Index (HBI) score < 4
6. Written informed consent obtained

Patient with Ulcerative Colitis

1. Aged ≥18 years old
2. Have a confirmed diagnosis of ulcerative colitis according to established clinical, endoscopic and histologic criteria
3. History of at least one flare with symptoms that required intervention within 24 months before screening
4. On stable regimen of 5-ASA for at least 3 months
5. In clinical remission for at least 3 months defined as partial Mayo score ≤ 1
6. Written informed consent obtained

Exclusion Criteria:

1. Previous bowel surgery /stoma
2. On anti-TNF therapy
3. Malignant disease within 5 years
4. Use of probiotics, prebiotics or antibiotics in past 3 months
5. Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients who visit Prince of Wales Hospital in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-01-28 (Estimated); Study Completion 2021-01-28 (Estimated)

PRIMARY OUTCOMES:
Clinical relapse for CD patients | 2 years
  Defined as worsening of the symptoms, accompanied by HBI score of ≥ 8 points for CD and require a change in therapy.
Clinical relapse for UC patients | 2 years
  Defined as partial Mayo score of ≥ 5 points for UC and require a change in therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, Prof, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Garcia-Sanchez V, Iglesias-Flores E, Gonzalez R, Gisbert JP, Gallardo-Valverde JM, Gonzalez-Galilea A, Naranjo-Rodriguez A, de Dios-Vega JF, Muntane J, Gomez-Camacho F. Does fecal calprotectin predict relapse in patients with Crohn's disease and ulcerative colitis? J Crohns Colitis. 2010 Jun;4(2):144-52. doi: 10.1016/j.crohns.2009.09.008. Epub 2009 Dec 2. PMID 21122498
- [Background] Hanaway P, Roseth A. Inflammatory biomarkers predict relapse in IBD. Gut. 2005 Sep;54(9):1346-7. doi: 10.1136/gut.2005.070615. No abstract available. PMID 16099806
- [Background] Sartor RB, Wu GD. Roles for Intestinal Bacteria, Viruses, and Fungi in Pathogenesis of Inflammatory Bowel Diseases and Therapeutic Approaches. Gastroenterology. 2017 Feb;152(2):327-339.e4. doi: 10.1053/j.gastro.2016.10.012. Epub 2016 Oct 18. PMID 27769810
- [Background] McIlroy J, Ianiro G, Mukhopadhya I, Hansen R, Hold GL. Review article: the gut microbiome in inflammatory bowel disease-avenues for microbial management. Aliment Pharmacol Ther. 2018 Jan;47(1):26-42. doi: 10.1111/apt.14384. Epub 2017 Oct 16. PMID 29034981
- [Background] Pascal V, Pozuelo M, Borruel N, Casellas F, Campos D, Santiago A, Martinez X, Varela E, Sarrabayrouse G, Machiels K, Vermeire S, Sokol H, Guarner F, Manichanh C. A microbial signature for Crohn's disease. Gut. 2017 May;66(5):813-822. doi: 10.1136/gutjnl-2016-313235. Epub 2017 Feb 7. PMID 28179361
- [Background] D'Haens G, Ferrante M, Vermeire S, Baert F, Noman M, Moortgat L, Geens P, Iwens D, Aerden I, Van Assche G, Van Olmen G, Rutgeerts P. Fecal calprotectin is a surrogate marker for endoscopic lesions in inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2218-24. doi: 10.1002/ibd.22917. Epub 2012 Feb 16. PMID 22344983